CLINICAL TRIAL: NCT00726349
Title: Transfusion Requirements in Orthopedic Surgery (Phase 2): A Prospective Observational Evaluation of the Optimal Transfusion Trigger.
Brief Title: Transfusion Requirements in Orthopedic Surgery (PHASE 2)
Acronym: TRIOS
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Dr Jean-François Hardy, Centre de recherche du CHUM (CRCHUM)
Other Study IDs: HD 06.084
Record Dates: First submitted 2008-07-29; First posted 2008-07-31 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2011-05

CONDITIONS: Total Hip or Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients undergoing isolated elective total hip or knee arthroplasty (primary or revision surgery for a non-malignant condition), aged 60 years or older and able to walk prior to surgery.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study.

SUMMARY:
The objective of our research program is to determine the transfusion threshold required to maximize functional recovery after major orthopedic surgery (total hip/knee replacement) in these, most often, elderly patient with serious comorbidities.

Hypothesis: we hypothesize that a threshold hemoglobin concentration exists below which functional recovery becomes difficult, even if the vital prognosis of patients is not impaired.

DETAILED DESCRIPTION:
Anemia is frequent after a surgical procedure. Postoperative anemia is associated with an increased incidence of transfusions and, probably, with an increased incidence of morbidity and mortality. However, the majority of studies evaluating the consequences of postoperative anemia are retrospective and, since anemic patients were transfused, they are unable to distinguish between the effects of anemia per se and those of transfusion. In orthopedic surgery, only two randomized controlled trials (RCT) have attempted to determine the benefits of transfusions in this patient population. The first evaluated the benefits of allogeneic transfusions in patients undergoing surgery for a fractured hip while the second evaluated autologous transfusions in patients undergoing total knee replacement. The small number of patients included in both studies did not allow definitive conclusions on the benefits (or lack thereof) of transfusions in orthopedic surgery.

Traditionally, a transfusion trigger of 100 g/L has been recommended in the postoperative period, especially in older patients and in those with serious comorbidities. In the Transfusion Requirements in Critical Care trial, a much lower transfusion threshold (70 g/L) was adopted in the group of patients in whom transfusions were restricted. This prospective randomized trial that included 838 patients, is, to this day, the most important in the field and generated unexpected results. Serious morbidity (cardiac and respiratory in particular) and mortality were not increased by the adoption of a low transfusion trigger while the number of transfusions was decreased significantly.

On the other hand, it is common to observe fatigue, decreased exercise capacity and muscle strength, and impaired performance of activities of daily life in the presence of anemia, especially when the hemoglobin concentration decreases below 90 - 100 g/L. In orthopedic surgery, a decrease in "postoperative vigor" can prevent patients from undertaking the rehabilitation program required to improve functional recovery after hip fracture repair.

The objective of our research program is to determine the transfusion threshold required to maximize functional recovery after major orthopedic surgery (total hip/knee replacement) in these, most often, elderly patient with serious comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing isolated elective total hip or knee arthroplasty (primary or revision surgery for a non-malignant condition), aged 60 years or older and able to walk prior to surgery.

Exclusion Criteria:

* Since this an observational study, all patients conforming to inclusion criteria will be included.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing isolated elective total hip or knee arthroplasty (primary or revision surgery for a non-malignant condition), aged 60 years or older and able to walk prior to surgery.
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2008-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Distance walked in 6 minutes after the operation. This is a simple, objective and reliable measure of functional recovery. | 4 to 6 days after surgery

SECONDARY OUTCOMES:
Fatigue, dizziness, difficulty to mobilize, difficulty/inability to participate in physiotherapy, prolonged hospital stay, major adverse events (especially cardiac, respiratory, neurological or infectious), death, impact of anemia on quality of life. | up to 4-6 days after surgery
Long-term functional status | 12 months following surgery
Long-term quality of life | 12 months following surgery
Long-term complications related to perioperative anemia | 12 months following surgery
  Evidence of myocardial ischemia, respiratory tract infections or other majors infections

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Hardy, MD, FRCPC, Principal Investigator — Centre Hospitalier Université Montréal
Locations (1):
- CHUM-Hôpital Notre-Dame, Montreal, Quebec, Canada